CLINICAL TRIAL: NCT00425581
Title: N-Terminal Pro-B-Type and Cardiac Troponin T Levels for Monitoring Effectiveness of Treatment in Very Low Birth Weight Infants With Hemodynamic Instability
Brief Title: N-Terminal Pro-B-Type Natriuretic Peptide and Troponin Levels as Markers of Hemodynamic Stability in Very Low Birth Weight Infants During the First Days of Life
Status: Withdrawn | Type: Observational
Why Stopped: Did not receive budget needed.
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Iris Morag, Sheba Medical Center
Other Study IDs: SHEBA-06-4255-IM-CTIL
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Hypotension; Very Low Birth Weight Infants; Ventricular Dysfunction; Prematurity
Keywords: N-terminal pro-BNP,; Cardiac Troponin-T,; Very low birth weight infants; hemodynamic instability; myocardial dysfunction
MeSH Terms: conditions — Hypotension; Ventricular Dysfunction; Premature Birth; Cardiomyopathy, Familial Restrictive, 3

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to test the hypothesis that there is an association between the hemodynamic status and the serum levels of NT-proBNP and cTnT in prematurely born infants. We would also evaluate the hypothesis that there is an association between the level of these proteins in the serum and the short and long term morbidity.

DETAILED DESCRIPTION:
NT-proBNP is a member of the natriuretic hormone family which plays an important role in regulation of extracellular fluid volume and blood pressure.It is secreted from the cardiac ventricle myocytes in response to myocardial stress. This hormone serves as a marker of ventricular dysfunction in adults but its role in newborns and especially preterm infants has not been well studied yet. Following birth of a healthy infant there is a surge in NT-proBNP levels which is then followed by a rapid decrease. One explanation for this surge is the transition in hemodynamics from fetal circulation into postnatal one. Few studies conducted in this area have shown association between NT-proBNP level and patency of ductus arteriosus and with respiratory distress syndrome of the newborn. Cardiac troponin T (cTnT)is a specific cardiac protein which serves as a specific indicator of cardiac damage in adults, it is usually not detected at birth but following myocardial injury its serum levels will slowly rise and generally will not be detectable until at least 4 hours after onset of injury. There is no "gold standard" test for diagnosis of hemodynamic instability in very low birth weight infants. Myocardial dysfunction is thought to be the major cause for this condition in VLBW population. Since this condition is associated with severe short and long term morbidity early recognition and specific treatment may be detrimental. We hypothesized that NT-proBNP and cTnT levels may serve as a more accurate markers for diagnosis, monitoring, and outcome prediction in VLBW infants during the first days of life, than the methods we currently use (blood pressure, urine output etc.)

ELIGIBILITY:
Inclusion Criteria:

* VLBW infants born at Sheba medical Center

Exclusion Criteria:

* known cardiac or chromosomal anomaly

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Iris Morag, MD, Principal Investigator — Sheba Medical Center

REFERENCES:
- [Background] Bar-Oz B, Lev-Sagie A, Arad I, Salpeter L, Nir A. N-terminal pro-B-type natriuretic peptide concentrations in mothers just before delivery, in cord blood, and in newborns. Clin Chem. 2005 May;51(5):926-7. doi: 10.1373/clinchem.2005.048892. No abstract available. PMID 15855678
- [Background] Nasser N, Bar-Oz B, Nir A. Natriuretic peptides and heart disease in infants and children. J Pediatr. 2005 Aug;147(2):248-53. doi: 10.1016/j.jpeds.2005.03.051. No abstract available. PMID 16126059
- [Background] Makikallio K, Vuolteenaho O, Jouppila P, Rasanen J. Ultrasonographic and biochemical markers of human fetal cardiac dysfunction in placental insufficiency. Circulation. 2002 Apr 30;105(17):2058-63. doi: 10.1161/01.cir.0000015505.24187.fa. PMID 11980685
- [Background] Cowie MR, Mendez GF. BNP and congestive heart failure. Prog Cardiovasc Dis. 2002 Jan-Feb;44(4):293-321. doi: 10.1053/pcad.2002.24599. PMID 12007084
- [Background] Puddy VF, Amirmansour C, Williams AF, Singer DR. Plasma brain natriuretic peptide as a predictor of haemodynamically significant patent ductus arteriosus in preterm infants. Clin Sci (Lond). 2002 Jul;103(1):75-7. doi: 10.1042/cs1030075. PMID 12095406